CLINICAL TRIAL: NCT03710057
Title: A Post-Marketing, Prospective, Observational Program: Effect of Ivabradrine in Lowering Heart Rate and Quality of Life in Chronic Heart Failure Patients
Brief Title: Effect of Ivabradine in Lowering Heart Rate and Quality of Life in Chronic Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Getz Pharma (Industry)
Responsible Party: Principal Investigator, Dr. Fawad Farooq, Assistant Professor, Consultant Cardiologist, National Institute of Cardiovascular Diseases, Pakistan
Other Study IDs: GTZ-CVD-001
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Chronic Heart Failure
Keywords: Ivabradine; Heart Rate; Health Related Quality of Life; Safety; Chronic Heart Failure Patient
MeSH Terms: interventions — Ivabradine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ivabradine — A prospective, post-marketing observational study was conducted in National Institute of cardiovascular disease, Karachi-Pakistan. Total 50 patients were advised to take 5 mg Ivabradine (SIVAB) twice daily for 8 weeks.

SUMMARY:
Elevated Heart rate (HR) (≥ 70 bpm) is one of the contributing factors in increasing the burden of hospitalization among Heart Failure patient. Ivabradine is a novel, selective and specific in inhibiting a Funny current in sinoatrial node Node and approved as an alternative therapy for Chronic Heart Failure (CHF) patients. CHF patients when treated with Ivabradine reported 39%, and 30% reduction in mortality and hospitalization rate respectively. Patient were treated with Ivabradine 5mg twice daily to determine its effect in lowering Heart rate and the Quality of Life (QOL) in Chronic Heart Failure patients

DETAILED DESCRIPTION:
A prospective, post-marketing observational study was conducted in 50 chronic heart failure patients with age 30-70yrs of NYHA Class II and prescribed 5 mg Ivabradine twice daily. Heart rate was evaluated through ECG & quality of life was measured by a validated questionnaire EuroQol-5 Dimension 3 level version (EQ-5D-3L). Baseline demographic includes age, gender, height, weight, Body Mass Index, temperature, blood pressure and respiratory rate were recorded and patients were followed at week 4 and week 8. Safety and tolerability was assessed by adverse drug reaction (ADR) monitoring. Results were analyzed by statistical software SPSS version 20.0.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Known case of Chronic Heart Failure (New York Heart Association (NYHA) functional class II to III)
* Clinically stability (at least for 4 weeks)
* Resting heart rate of more than 70 beats/ min (bpm) as assessed from the 12-lead electrocardiogram.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Resting heart rate below 70 beats per minute prior to treatment
* Cardiogenic shock
* Acute myocardial infarction
* Severe hypotension (< 90/50 mmHg)
* Severe hepatic insufficiency
* Sick sinus syndrome
* Sino-atrial block
* Unstable or acute heart failure
* Pacemaker dependent (heart rate imposed exclusively by the pacemaker)
* Unstable angina
* Atrioventricular Block of 3rd degree
* The combination with a strong cytochrome P450 3A4 inhibitors such as azole antifungals (ketoconazole, itraconazole), macrolide antibiotics (clarithromycin, erythromycin, telithromycin), HIV protease inhibitors (nelfinavir, ritonavir) and nefazodone
* The combination with verapamil or diltiazem which are moderate CYP3A4 inhibitors with heart rate reducing properties.
* Pregnancy, lactation and women of child-bearing potential not using appropriate contraceptive measures

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was included male or female patients with Chronic Heart Failure (CHF). Diagnosis of CHF as per Boston Criteria for Diagnosing Heart failure and the New York Heart Association (NYHA) functional class II to III classification and rest on the based on the medical judgment of the investigator after review of subject's medical history, results of routine screening physical and general examination and routine laboratory investigations.
  Patients' written authorization was used to obtain patients' data. However, patient data secrecy was followed by ICH GCP requirements.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Mean difference of Heart Rate | at 4 week and 8 week
  The primary end-point was the overall response rate of patients to Ivabradine in achieving HR <70 Bpm

SECONDARY OUTCOMES:
Percentage of problems reported in EQ-5D descriptive system | at 4 week and 8 week
  Quality of Life was determined through validated questionnaire EQ-5D-3L. It also assesses five dimensions of HR quality of life (HRQoL): mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension is measured one to three levels i.e 1, 2, 3. Where level 2 & 3 indicates 'problem' and level 1 denotes to 'no problem'.
Median score of EQ-5D visual analogue scale | at 4 week and 8 week
  The EQ-5D registers the self-rated health status of the respondent on the vertically visual analogue scale (EQ-5D VAS) from 0 to 100 where 100 indicates 'Best imaginable health' and 0 is said to be a 'Worst imagine health state'.

OTHER OUTCOMES:
Percentage of Reported Adverse Drug Reactions | upto 8 weeks
  The pre-defined secondary outcome was to determine Safety and tolerability by monitoring adverse drug reactions.